CLINICAL TRIAL: NCT04429815
Title: Impact of Smoking and Nicotine on the Risk of Being Infected With COVID-19
Acronym: MAGIC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01681-38
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active smokers.: Active smokers since October 2019.
  Interventions: Diagnostic Test: Serological test for COVID-19.
- Smokers undergoing smoking cessation: Smokers undergoing smoking cessation and taking nicotine substitutes on a regular basis since October 2019.
  Interventions: Diagnostic Test: Serological test for COVID-19.
- Non-smoking.: Person who's never smoked before.
  Interventions: Diagnostic Test: Serological test for COVID-19.

INTERVENTIONS:
Diagnostic Test: Serological test for COVID-19. — Serological test for COVID-19 performed as part of standard of care.

SUMMARY:
Several studies have shown that smokers have a higher risk of developing a severe form of COVID-19 once a person has been infected. This is explained by the damage caused by smoking at the bronchopulmonary level and an overexpression of some coronavirus receptors at the pulmonary level when exposed to tobacco. In contrast, recent data indicate that smokers are proportionally less infected with the COVID-19 virus since all available cohort data from around the world show a very low rate of smokers among COVID-19 infected subjects. The mechanisms at the origin of this protective effect are not known. All of these data lead us to question the real role of nicotine in the protective effect of tobacco observed in the general population against infection by the COVID-19 virus.

The objectives are :

* To show that subjects taking nicotine substitutes as part of a smoking cessation program are less infected with COVID-19 than non-smokers.
* To show that active smokers are less infected with COVID-19 than non-smokers.
* To compare the percentage of positive serological tests in subjects taking nicotine substitutes to the percentage of positive serological tests in active smokers.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Subject who will require a serological test for COVID-19 virus as part of standard of care.
* Group 1: Active smoker since October 2019
* Group 2: Smoker undergoing smoking cessation and taking nicotine substitutes on a regular basis since October 2019
* Group 3: Non-smoker

Exclusion Criteria:

* Inpatient subject
* Subjects with a chronic serious pathology modifying the risk of exposure to COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects (smokers, smokers undergoing smoking cessation, non-smokers) who will require a serological test for COVID-19 as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a positive serological test for COVID-19. | 1 day
  Percentage of patients with a positive serological test for COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rabaud, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No